CLINICAL TRIAL: NCT03937882
Title: A Multi-Center, Randomized, Double Masked, Placebo Controlled Clinical Study to Assess the Safety and Efficacy of RGN-259 Ophthalmic Solutions for the Treatment of Dry Eye (ARISE-3)
Brief Title: Assessment of the Safety and Efficacy of RGN-259 Ophthalmic Solutions for Dry Eye Syndrome: ARISE-3
Acronym: ARISE-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ReGenTree, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGN-259/19-110-0002
Record Dates: First submitted 2019-05-01; First posted 2019-05-06 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye Syndromes; Dry Eye
Keywords: Dry Eye; Dry Eye Syndrome; DES
MeSH Terms: conditions — Dry Eye Syndromes | interventions — thymosin beta(4)

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 1:1 ratio RGN-259 to placebo ophthalmic solution.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects, investigators, and study personnel involved with the conduct of the study will be masked with regard to treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RGN-259 (Experimental): RGN-259: It is a preservative-free, sterile eye drop solution containing Thymosin beta 4
  Interventions: Drug: RGN-259
- Placebo (Placebo Comparator): It is composed of the same excipients as RGN-259 but does not contain Thymosin beta 4
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RGN-259 — A preservative-free, sterile eye drop solution containing Thymosin beta 4 for direct instillation into each eye, four times a day (QID) for 14 days
  Other Names: Tβ4; Thymosin Beta 4
  Arms: RGN-259
Drug: Placebo — It is composed of the same excipients as RGN-259 but does not contain Thymosin beta 4
  Other Names: Vehicle Control
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the safety and efficacy of RGN-259 Ophthalmic Solution to placebo for the treatment of the signs and symptoms of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a subject reported history of dry eye for at least 6 months;
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months

Exclusion Criteria:

* Have any clinically significant slit-lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction (MGD), lid margin inflammation or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
* Have an uncontrolled systemic disease;
* Be a woman who is pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2020-11-08 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Corneal staining | 15 days after first dosing
  Mean change from baseline to Day 15 of Inferior Corneal Fluorescein Staining
Ocular Discomfort 6-point (0=none, 5=worst) scale | 15 days after first dosing
  Mean change from baseline to Day 15 of Ocular Discomfort severity

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Eye Research Foundation, Newport Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Dovilan Wyatt MD, LLC, Chicago, Illinois
  - Whitson Vision, Indianapolis, Indiana
  - Midwest Cornea Associates, LLC, Indianapolis, Indiana
  - The Eye Care Institute, Louisville, Kentucky
  - Andover Eye Associates, Andover, Massachusetts
  - Andover Eye Associates, Raynham, Massachusetts
  - Center For Sight, Henderson, Nevada
  - Oculus Research, Inc. at the Eye Care Center, Raleigh, North Carolina
  - Visual Eyes Optometric, Shelby, North Carolina
  - Bergstrom Eye Research, LLC, Fargo, North Dakota
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Andover Eye Associates, Warwick, Rhode Island
  - Total Eye Care, P.A., Memphis, Tennessee
  - Texan Eye/Keystone Research, Austin, Texas
  - Mountain View Eye Center, Layton, Utah
  - Country Hills Eye Center, Ogden, Utah
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No